CLINICAL TRIAL: NCT01392092
Title: Effects of N-acetylcysteine on Brain Chemistry and Behavior in Cocaine Abusers
Brief Title: Effects of N-acetylcysteine on Brain Chemistry and Behavior in Cocaine Abusers (NAC)
Acronym: NAC
Status: Completed | Type: Observational
Sponsor: Wayne State University (Other)
Responsible Party: Principal Investigator, Mark Greenwald, PhD, Principal Investigator, Wayne State University
Other Study IDs: NAC-1
Record Dates: First submitted 2011-07-11; First posted 2011-07-12 (Estimated); Last update posted 2018-04-05 (Actual); Status verified 2018-04

CONDITIONS: Cocaine Abuse or Dependence; Cocaine Related Disorders
Keywords: Contingency Management; Drug Self-Administration
MeSH Terms: conditions — Cocaine-Related Disorders

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
N-acetylcysteine (NAC) is a medication that the Food and Drug Administration (FDA) has approved for several medical uses, such as dissolving mucus in patients with breathing problems, treating overdose from acetaminophen (Tylenol), and protecting the kidneys from toxic substances.

Some recent studies suggest that NAC could be useful in the treatment of other disorders including addictions. One purpose of this study is to determine whether NAC alters the level of brain glutamate (a chemical that excites brain cells). The other main purpose is to determine whether NAC affects how much cocaine people use.

DETAILED DESCRIPTION:
Inpatient Phase: Participants will live on an inpatient research unit at least 2 consecutive nights and possibly up to 20 consecutive nights. Participants cannot have visitors and will not be allowed to leave the inpatient unit (except with a staff escort) unless they drop out of the study. We will collect daily urine samples to make sure participants are not using any drugs except those in the study. In addition, each morning, afternoon and evening participants will receive a capsule containing placebo (a blank) or different doses of N-acetylcysteine.

Participants will take part in multiple trials (up to 9 sessions) where they will be given a standard amount of powder (identified as Drug A or Drug B) to inhale through a straw into their nose. The powder will contain placebo (a powder containing no drug) or different doses of cocaine. We will measure how participants are feeling using questionnaires and we will record vital signs-including breathing rate, blood oxygen level, heart rate, and blood pressure.

Participants will also be asked to perform a 3-hour computer task that allows them to work for Drug A, Drug B, or money. At the end of the computer task participants will receive the amount of drug they earned and a receipt for the amount of money they earned.

On each Monday of the inpatient stay, participants will be escorted to Harper Hospital for a special type of magnetic resonance imaging (MRI) scan, known as magnetic resonance spectroscopy (MRS). This is a non-invasive way to study brain chemistry. Participants will take part in a total of two (2) MRI scans. The total length of each brain scan will be about 2 hours.

Additionally on each Monday of the inpatient stay we will test the sensitivity of the participants brain to magnetic stimulation. A small magnet will be placed on top of the head so that a small electrical current is generated inside the brain. This procedure is called transcranial magnetic stimulation (TMS). We will stimulate the part of the brain that controls finger movement. Three recording electrodes (metal sensors like those used for EKG) will be placed on the right thumb and index fingers. We will measure the effects of different amounts of magnetic stimulation on the muscle activity of the thumb and index fingers (as seen on a computer screen). We will also ask participants to push a lever with their finger during parts of the procedure. These tasks will last about 2 hours.

To complete the study, a minimum stay of 16 inpatient nights is required. The maximum stay is 20 inpatient nights.

ELIGIBILITY:
Inclusion Criteria:

* Male and female volunteers (18-55 years of age)
* Must meet DSM-IV criteria for current Cocaine Abuse or Dependence and wish to participate in research.
* Positive urine test for cocaine.
* Candidates must be in good health to be eligible.
* All candidates must receive routine medical (history and physical) exam with standard laboratory tests (complete blood chemistry, urinalysis, urine pregnancy test for females, tuberculin screening), and 12-lead ECG at the initial screening visit.

Exclusion Criteria:

* Serious psychiatric illness (e.g. psychosis, bipolar, suicide attempts, major depression that is not substance-induced).
* Substance use disorder other than cocaine abuse or dependence, nicotine dependence, alcohol abuse, sedative abuse or marijuana abuse.
* Neurological diseases (e.g. stroke, seizures); cardiovascular problems (e.g. myocardial infarction, angina, systolic BP >160 or <95 mmHg, diastolic BP >95 mmHg, or clinically abnormal ECG); pulmonary diseases (e.g. asthma, TB); systemic diseases (e.g. hepatitis, autoimmune diseases).
* Cognitive impairment.
* Exposed in past 30 days to medications that would increase study risk (e.g. toxicity to major organ systems, psychotropics, asthma inhalers, or interactions with study drugs).
* Pregnant (urine HCG), lactating (self-report), or if heterosexually active and not using (self-report) medically approved birth control measures (oral or depot contraceptives, IUD, condom/foam, sterilization, tubal ligation).
* Seeking treatment or being treated for a substance use disorder.
* Metal objects in body (e.g. metal plates, part of a bullet from a gunshot wound, or a catheter).

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Cocaine abusing or dependent research volunteers
Sampling Method: Non-Probability Sample
Enrollment: 16 (Actual)
Dates: Start 2011-07; Primary Completion 2017-06 (Actual); Study Completion 2017-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mark Greenwald, PhD, Principal Investigator — Wayne State University
Locations (1):
- Wayne State University, Detroit, Michigan, United States